CLINICAL TRIAL: NCT05657158
Title: Retrospective Analysis of Imaging and Clinical Features From Patients Treated With Brolucizumab in Post-marketing Setting With Reports of Intraocular Inflammation and/or Retinal Vascular Occlusion
Brief Title: Analysis of Imaging Features From Patients Treated With Brolucizumab in the Post-marketing Setting With Reports of Retinal Vasculitis and/or Retinal Vascular Occlusion
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258A2404
Record Dates: First submitted 2022-11-16; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Intraocular Inflammation; Retinal Vascular Occlusion
Keywords: Brolucizumab; Neovascular age-related macular degeneration; occlusive retinal vasculitis; retinal vasculitis; RV; retinal vascular occlusion; RO; ocular images
MeSH Terms: conditions — Uveitis; Retinal Vasculitis | interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Brolucizumab: brolucizumab in routine clinical practice
  Interventions: Other: Brolucizumab

INTERVENTIONS:
Other: Brolucizumab — Participants with cases of RV and/or RO reported to Novartis Patient Safety following brolucizumab use in routine clinical practice for which images were provided to Novartis and read by the Reading Centre were included

SUMMARY:
This non-interventional descriptive study was undertaken to better understand the most common imaging features associated with inflammation arising in the post-marketing setting when brolucizumab was prescribed in routine clinical practice.

DETAILED DESCRIPTION:
The purpose of this retrospective study analysis was to better characterize the risk of inflammatory events arising from use of brolucizumab in routine clinical practice through analysis of independently reviewed ocular imaging data obtained from cases with reports of intraocular inflammation (IOI), retinal vasculitis (RV) and/or Retinal vascular occlusion (RO) and to provide a description of these features.

Whenever an AE report pertaining to RV and/or RO was reported to Novartis Patient Safety, a follow-up check list (targeted follow-up checklists [TFUs]) was sent by Novartis to the reporter. The reporter was encouraged to share all available images obtained as part of clinical practice, irrespective of the timing or event (i.e. images before, during, and after event could be provided). The focus and main efforts of this data collection was on adverse events of RV and/or RO; for other IOI only events, the images were not actively requested in the case documentation process, however in some cases these were spontaneously reported by the reporter.

All images obtained from Feb 2020 up to 31 Jan 2021 were reviewed in a standardized manner by an external reading center. Dedicated grading lists were developed for each of the image modalities: Fluorescein Angiography (FA), Fundus Photography (FP), Indocyanine Green Angiography (ICGA), Optical Coherence Tomography (OCT), and OCT Angiography (OCT-A).

ELIGIBILITY:
Inclusion Criteria:

* participants with cases of RV and/or RO reported to Novartis Patient Safety following brolucizumab use in routine clinical practice for which images were provided to Novartis and read by the Reading Centre

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As this study used secondary data from Novartis Patient Safety database, there was no specified set of subject population in this study and all cases with event of interest and available images were retrieved.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-01-04 (Actual)

PRIMARY OUTCOMES:
Eye case classification based on imaging data | throughout the study period of 5 months
  Eye case classification based on imaging data is provided:
  * IOI: intraocular inflammation (posterior segment only)
  * RV: Retinal vasculitis
  * RO: Retinal vascular occlusion
  * Not assessable: image quality concerns prevented grading
  * None: no imaging features of IOI, RV, or RO
Number of eye cases by anatomical location and sub-location | throughout the study period of 5 months
  Number of eye cases by anatomical location and sub-location is provided:
  * Retina: Vascular and general)
  * Vitreous
  * Choroid
  * Optic nerve
Number of eye cases by occlusion type by reading center eye case classification | throughout the study period of 5 months
  Occlusion type by reading center eye case classification is provided:
  * Central
  * Branch
  * Peripheral
Number of eye cases by Anatomical location in relation to macula | throughout the study period of 5 months
  Number of eye cases by Anatomical location in relation to macula is provided:
Number of eye cases by extent of involvement of the retinal arterial and vein occlusion | throughout the study period of 5 months
  Number of eye cases by Extent of involvement of the retinal arterial and vein occlusion is provided
Number of eye cases by grading variables per imaging modality by reading center eye case classification | throughout the study period of 5 months
  Number of eye cases by grading variables per imaging modality by reading center eye case classification is provided

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative center, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No